CLINICAL TRIAL: NCT01494818
Title: Evaluation of the Effects of Clear Care/AOSEPT Plus Hydrogen Peroxide Solution on the Eyelid Tissues - Part II: Comparative Evaluation With RENU MPS Over 3 Months of Wear
Brief Title: Evaluation of Marketed Contact Lens Disinfectant Systems on Eyelid Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ID 10-59 / M-11-02
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-07

CONDITIONS: Contact Lens Care
Keywords: Contact lenses; Contact lens solutions
MeSH Terms: interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLEAR CARE/AOSEPT Plus (Experimental): Hydrogen peroxide-based contact lens care system used per manufacturer's instructions
  Interventions: Device: Hydrogen peroxide-based contact lens care system; Device: Soft contact lenses
- ReNu MultiPlus (Active Comparator): PHMB-containing contact lens solution used per manufacturer's instructions
  Interventions: Device: PHMB-containing contact lens solution; Device: Soft contact lenses

INTERVENTIONS:
Device: Hydrogen peroxide-based contact lens care system
  Other Names: CLEAR CARE®/AOSEPT Plus
  Arms: CLEAR CARE/AOSEPT Plus
Device: PHMB-containing contact lens solution
  Other Names: ReNu® MultiPlus Multi-Purpose solution
  Arms: ReNu MultiPlus
Device: Soft contact lenses — Contact lenses identical to habitual prescription worn per usual replacement regimen

SUMMARY:
The purpose of this study was to assess and compare the effect of the repeated usage of two different contact lens care systems (one hydrogen peroxide-based cleaning and disinfecting system, and one polyaminopropyl biguanide (PHMB)-containing multipurpose system) with silicone hydrogel contact lenses worn on a daily wear basis for three months. The specific aspect of interest was the effect on the ocular tissue, in particular the eyelids and their associations with the contact lens surface wettability and surface contamination.

DETAILED DESCRIPTION:
The subjects attended the enrollment visit having worn their habitual silicone hydrogel contact lenses for at least six hours on the day of the visit. The enrollment visit was scheduled so that the subjects' habitual lenses were at least 14 ± 3 days old for the subjects replacing their lenses bi-weekly and at least 30 ± 5 days old for those replacing their lenses monthly.

ELIGIBILITY:
Inclusion Criteria:

* Read and understand Participant Information Sheet;
* Read, sign, and date Informed Consent;
* Successfully wearing silicone hydrogel contact lenses under a frequent replacement (biweekly or monthly) daily wear modality;
* Using a PHMB-containing multipurpose contact lens solution;
* Symptomatic, as specified in protocol;
* Best corrected visual acuity of 6/9 or better in each eye;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any known sensitivity or intolerance to the contact lenses or len care products to be used;
* Systemic disease/medication which might interfere with contact lens wear or produce dry eye side effects;
* Ocular allergies or ocular disease which might interfere with contact lens wear;
* Use of any concomitant topical ocular medications during the study period;
* Participation in an investigational drug or device study within 30 days of entering the study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Guillon, PhD, FCOptom, FAAO, CCTI, Principal Investigator — OTG Research & Consultancy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one study center located in the United Kingdom.
Pre-assignment Details: Of the 79 participants enrolled in the study, 1 participant exited the study between enrollment and product dispensing due to nonavailability. This reporting group includes all enrolled and dispensed participants.
Groups:
- CLEAR CARE/AOSEPT Plus: Hydrogen peroxide-based contact lens care system used with silicone hydrogel contact lenses per manufacturer's instructions for 3 months
- ReNu MultiPlus: PHMB-containing contact lens solution used with silicone hydrogel contact lenses per manufacturer's instructions for 3 months
Period: Overall Study
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Started | 39 | 39
Completed | 37 | 37
Not Completed | 2 | 2
Not completed — Relocation | 1 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled and dispensed participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus | Total
Number analyzed (Participants) | 37 | 37 | 74
Age Continuous [Mean (Standard Deviation); unit: years] | 34.8 (9.8) | 35.5 (10.5) | 35.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximum Papillae
Description: Eyelid papillae (bumps on the inner eyelid) were recorded separately for three zones of the upper lid and overall for the lower lid on a 5-point forced choice scale (0 = None; 1 = Slight (diffuse papillae); 2 = Mild (diffuse & tufts papillae); 3 = Moderate (moderate & tufts papillae); 4 = Severe (giant papillae). The maximum value represents the worse grade in any zone. Both eyes were included in the model for analysis.
Time Frame: Baseline, Month 3
Population: All enrolled and dispensed participants who completed the study as per protocol
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 37 | 37
Units on a scale
  Baseline (habitual contact lenses and care system) | 2.0 [0 to 4] | 2.0 [0 to 3]
  Month 3 | 2.0 [0 to 3] | 2.0 [0 to 3]

2. Primary Outcome: Maximum Eyelid Hyperaemia
Description: Eyelid hyperaemia (redness) was recorded separately for three zones of the upper lid and overall for the lower lid on a 5-point forced choice scale (0 = Clear; 1 = Slight redness; 2 = Mild redness; 3 = Moderate redness; 4 = Severe redness). The maximum value represents the worst grade in any zone. Both eyes were included in the model for analysis.
Time Frame: Baseline, Month 3
Population: All enrolled and dispensed participants who completed the study as per protocol
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 37 | 37
Units on a scale
  Baseline (habitual contact lenses and care system) | 2.0 [1 to 4] | 2.0 [1 to 4]
  Month 3 | 2.0 [1 to 3] | 2.0 [1 to 3]

3. Secondary Outcome: Median Non-Invasive Pre-Lens Tear Film Break Up Time (PL-NIBUT)
Description: The pre-lens tear film is the layer of tears located on top of the contact lens (i.e., between the eyelid and the contact lens). The time required for a dry spot to appear on the pre-lens surface after blinking is referred to as the pre-lens tear film break up time. PL-NIBUT was evaluated using a biomicroscope with a diffuse illumination source, i.e., Tearscope. A longer PL-NIBUT indicates a more stable tear film and greater on-eye lens wettability. Three PL-NIBUT measurements were recorded, and the median value was used for analysis. Both eyes were included in the model for analysis.
Time Frame: Baseline, Month 3
Population: All enrolled and dispensed participants who completed the study as per protocol
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 37 | 37
Seconds
  Baseline (habitual contact lenses and care system) | 4.05 (4.63) [0.90 to 32.00] | 5.08 (4.07) [1.20 to 16.60]
  Month 3 | 5.76 (4.50) [1.00 to 24.70] | 4.22 (2.12) [1.30 to 12.20]

4. Primary Outcome: Upper Lid Redness
Description: The contact lenses were removed and upper lid redness was objectively measured through digital images. The coverage of the palpebral surface by blood vessels is expressed as percentage of the total surface measured. Both eyes were included in the model for analysis.
Time Frame: Baseline, Month 3
Population: All enrolled and dispensed participants who completed the study as per protocol
Measure: Mean (Standard Deviation); unit: Percentage of total surface measured
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 37 | 37
Percentage of total surface measured
  Baseline (habitual contact lenses and care system) | 34.8 (6.8) | 34.9 (6.1)
  Month 3 | 35.2 (7.0) | 35.4 (5.8)

5. Primary Outcome: Change From Baseline in Upper Eyelid Margin Staining at Month 3
Description: The contact lens was removed and ophthalmic dye was instilled. Upper eyelid margin staining was objectively measured through digital images. The extent of true staining (i.e., the total area of lid margin covered by staining) was recorded. Both eyes were included in the model for analysis.
Time Frame: Baseline, Month 3
Population: All enrolled and dispensed participants who completed the study as per protocol
Measure: Mean (Standard Deviation); unit: square millimeters
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 37 | 37
square millimeters | -0.014 (3.905) | -0.754 (4.179)

6. Secondary Outcome: Protective Index
Description: A digital video recording was made of the interblink period. The percentage of area of the visible contact lens covered by the tear film was calculated (Protected Area). The Protective Index is defined as the average tear coverage over the whole interblink period. Both eyes were included in the model for analysis.
Time Frame: Baseline, Month 3
Population: All enrolled and dispensed participants who completed the study as per protocol
Measure: Mean (Standard Deviation); unit: Percent of visible contact lens surface
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 37 | 37
Percent of visible contact lens surface
  Baseline (habitual contact lenses and care system) | 95.9 (11.0) | 95.8 (10.2)
  Month 3 | 96.4 (10.0) | 97.8 (5.8)

7. Secondary Outcome: Median Front Lens Deposits
Description: Deposits present on the front surface of the lens were assessed with a biomicroscope while the lens was on eye. Deposits were rated on a 5-point forced choice scale (0 = none; 1 = slight; = mild; 3 = moderate; 4 = severe) in five lens zones. The median of the five zones was used for analysis. Both eyes were included in the model for analysis.
Time Frame: Baseline, Month 3
Population: All enrolled and dispensed participants who completed the study as per protocol
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 37 | 37
Units on a scale
  Baseline (habitual contact lenses and care system) | 0 [0 to 2] | 0 [0 to 1]
  Month 3 | 0 [0 to 0] | 0 [0 to 2]

8. Secondary Outcome: Total Lipid Uptake Per Lens
Description: The contact lens was aseptically removed from the eye. Lipids were extracted and analyzed using a proprietary High Performance Liquid Chromatography technique. A lower value would indicate a cleaner lens surface.
Time Frame: Baseline, Month 3
Population: All enrolled and dispensed participants who completed the study as per protocol
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 37 | 37
micrograms
  Baseline (habitual contact lenses and care system) | 38.95 (23.94) [4.121 to 95.504] | 36.44 (47.59) [4.150 to 97.875]
  Month 3 | 32.40 (24.53) | 34.20 (26.57)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. The safety population includes all participants exposed to test product.
Description: An adverse event was any untoward medical occurrence in a subject administered a test article, regardless of causal relationship with the treatment.
Arm/Group | CLEAR CARE/AOSEPT Plus | ReNu MultiPlus
Serious Adverse Events (participants affected / at risk) | 2/39 | 0/39
Other Adverse Events (participants affected / at risk) | 3/39 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLEAR CARE/AOSEPT Plus (N=39) | ReNu MultiPlus (N=39)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLEAR CARE/AOSEPT Plus (N=39) | ReNu MultiPlus (N=39)
Toxic reaction to solution (Eye disorders) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.